CLINICAL TRIAL: NCT00722254
Title: Reversible Secondary Myelofibrosis or Clonal Myeloproliferative Disorder
Status: Terminated | Type: Observational
Why Stopped: This study was stopped due to poor enrollment numbers
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 17806; 1P01CA108671-01A2 (NIH)
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Primary Myelofibrosis; Primary Pulmonary Hypertension; Secondary Myelofibrosis; Pulmonary Arterial Hypertension
Keywords: Myeloproliferative Disorder; Primary Myelofibrosis; Primary Pulmonary Hypertension; Secondary Myelofibrosis; Pulmonary Arterial Hypertension; Flolan; Clonality; CD34+ cells; Hematologic abnormalities
MeSH Terms: conditions — Primary Myelofibrosis; Familial Primary Pulmonary Hypertension; Pulmonary Arterial Hypertension; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PPH: Subjects diagnosed with primary pulmonary hypertension (PPH)
- Myelofibrosis: Subjects diagnosed with Primary or Secondary Myelofibrosis

SUMMARY:
To determine the prevalence of myelofibrosis in patients with primary pulmonary hypertension, and to discover if the fibrosis in these patients is primary (AMM) or secondary.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension: Pulmonary arterial hypertension (PAH) is a disease primarily affecting the small precapillary pulmonary vessels. It is characterized by sustained elevation of the pulmonary vascular resistance (PVR). Without therapy, right heart failure and death eventually occur. PAH occurs in an idiopathic form, primary pulmonary hypertension (PPH), and in association with other disorders such as connective tissue diseases or congenital heart disease (CHD). PAH remains a disease of unknown etiology. Until recently, prognosis for PAH was poor, with a median survival of less than 3 years.

Prostacyclin (PGI2) is the main product of arachidonic acid in all vascular endothelium. It is a potent vasodilator in all vascular beds. In addition, it is a potent endogenous inhibitor of platelet aggregation and smooth muscle growth. The prostacyclin receptor (IP) is located on a variety of cell types, enabling prostacyclin to exert a range of biologic actions by means of raising intracellular levels of cAMP through activation of adenylate cyclase. The stable, freeze-dried salt preparation of prostacyclin is known as epoprostenol and is available for IV administration under the brand name Flolan (Glaxo Wellcome, Research Triangle Park, N.C.). The first randomized clinical trial in PPH showed that epoprostenol improved quality of life, hemodynamics, exercise tolerance, and survival over a 12-week period. Epoprostenol has become the standard of care for patients with advanced PPH. Recently, chronic intravenous epoprostenol has been shown to be an effective therapy to improve long-term quality of life and survival in patients with PPH. Epoprostenol also improves hemodynamics, exercise capacity, and quality of life (but not survival) in PAH associated with CHD and connective tissue disease.

Side effects of epoprostenol infusion include rash, headache, jaw pain, leg pain, diarrhea, nausea, catheter infections, chest pain, anxiety dizziness, bradycardia, dyspnea, abdominal pain, musculoskeletal pain, tachycardia, flu-like symptoms, and anxiety/nervousness. Thrombocytopenia is commonly seen in patients with PPH treated with PG12. Occasionally, a decrease in other blood cell lines occurs leading to anemia or pancytopenia. Splenomegaly and hypersplenism are observed at times. While thrombocytopenia has been attributed to the antiplatelet effects of prostacyclin, the pathophysiology of pancytopenia is poorly understood. There are no studies that address thrombocytopenia and other hemopoietic abnormalities in people with pulmonary hypertension receiving epoprostenol. The possibility of myelofibrosis causing these hematologic abnormalities has not been investigated.

Primary myelofibrosis is a myeloproliferative disorder, characterized typically by pancytopenia, splenomegaly, a leukoerythroblastic blood smear, fibrosis on the bone marrow examination, and myeloid metaplasia. Like all myeloproliferative disorders, it is due to somatic mutation and clonal proliferation of hematopoietic progenitors. Fibrosis occurs secondary to cytokines secreted by malignant cells. These patients are symptomatic because of cytopenias. Bone marrow failure and transformation to acute myeloid leukemia is the major reason for mortality in these patients. Elevated blood levels of hematopoietic progenitors (identified by positivity for the CD34 antigen) are well documented and correlates with prognosis. Therefore two major identifying features of primary myelofibrosis as opposed to secondary fibrosis of the marrow are: 1) clonal hematopoiesis and 2) high CD 34 positive hematopoietic precursors.

We therefore hypothesize these two will be normal in patients with secondary myelofibrosis and help us distinguish the two entities.

Clonality Studies: Clonality is based on the principal of X-chromosome inactivation and thus, for clonality studies only females can be used as subjects. It is based on the principal that while female cells have two X-chromosomes, one is randomly inactivated during early embryonic development and thus female tissue is a mixture of cells expressing either paternal or maternal inherited x-chromosome genes. In the first step, DNA analysis will study 5 exonic polymorphisms for the X-chromosome genes which have previously been shown to be useful for these purposes. If any of the five loci is heterozygous then the subject is said to be informative for clonality. Studies which will proceed as follows: The fresh blood platelets and granulocytes will be isolated and the RNA isolated and used later for reverse transcription to cDNA which will then be analyzed for X-chromosome allelic usage ratio by single-stranded conformational polymorphisms (SSCP). If only one allele is expressed in platelets or granulocytes the patient is said to be clonal and favors a diagnosis of myeloproliferative disorder (such as AMM), while polyclonal blood (both X-chromosome alleles expressed in platelets and granulocytes) is compatible with secondary myelofibrosis.

A three-color direct immunofluorescent staining method will be used in the evaluation of CD34+ cells. In our preliminary experience we observed four Flolan treated patients with PPH who had splenomegaly, anemia and/or thrombocytopenia. All of these patients had severe marrow fibrosis. The purpose of this study is to determine whether the incidence of the bone marrow fibrosis in this patient population is primary or secondary, and whether a secondary effect is a fibrosis that would be expected to be transient and resolve after discontinuation of Flolan.

Participating subjects will Patients will undergo the following studies:

1. History and Physical examination
2. Peripheral blood smear
3. Bone marrow examination to determine the presence and severity of fibrosis. The bone marrow specimen taken for diagnostic purposes will be examined by three independent hematologists/hematopathologists in a masked fashion for the presence of fibrosis using routine methods.
4. Blood: 30 cc of blood will be collected for

   1. Clonality studies (female subjects only),
   2. CD34 quantitation.
   3. Further studies will be done to monitor the aberrant trafficking of hemopoietic stem cells, the adhesion molecules, and any disease related genes, such as JAK2V617F and cMPL, if indicated.
   4. The above studies will be repeated in patients undergoing lung transplants at 3 months, 6 months and 1 year after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. > 18 years of age
2. Signed Informed Consent
3. Subjects diagnosed with Primary Pulmonary Hypertension or Myelofibrosis (primary or secondary)

Exclusion Criteria:

1. Anyone not meeting the above inclusion criteria
2. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from primary pulmonary hypertension or myelofibrosis (primary or secondary)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of myelofibrosis in patients with primary pulmonary hypertension | After sample is obtained

SECONDARY OUTCOMES:
Discover if the fibrosis in patients with primary pulmonary hypertension is primary (AMM) or secondary. | After sample is obtained
Clonality | After sample is obtained

CONTACTS AND LOCATIONS:
Overall Officials: Josef T Prchal, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - VA Salt Lake City Health Care System, Salt Lake City, Utah

REFERENCES:
- [Background] Hoffman R, Prchal JT, Samuelson S, Ciurea SO, Rondelli D. Philadelphia chromosome-negative myeloproliferative disorders: biology and treatment. Biol Blood Marrow Transplant. 2007 Jan;13(1 Suppl 1):64-72. doi: 10.1016/j.bbmt.2006.11.003. PMID 17222772
- [Background] Chen GL, Liu E, Naidoo K, Popat U, Coetzer TL, Prchal JT. Idiopathic myelofibrosis without dacryocytes. Haematologica. 2006 Jun;91(6 Suppl):ECR29. PMID 16785132
- [Background] Popat U, Frost A, Liu E, Guan Y, Durette A, Reddy V, Prchal JT. High levels of circulating CD34 cells, dacrocytes, clonal hematopoiesis, and JAK2 mutation differentiate myelofibrosis with myeloid metaplasia from secondary myelofibrosis associated with pulmonary hypertension. Blood. 2006 May 1;107(9):3486-8. doi: 10.1182/blood-2005-08-3319. Epub 2006 Jan 17. PMID 16418333
- [Background] Popat U, Frost A, Liu E, May R, Bag R, Reddy V, Prchal JT. New onset of myelofibrosis in association with pulmonary arterial hypertension. Ann Intern Med. 2005 Sep 20;143(6):466-7. doi: 10.7326/0003-4819-143-6-200509200-00017. No abstract available. PMID 16172450
- [Background] Xu M, Bruno E, Chao J, Huang S, Finazzi G, Fruchtman SM, Popat U, Prchal JT, Barosi G, Hoffman R; MPD Research Consortium. Constitutive mobilization of CD34+ cells into the peripheral blood in idiopathic myelofibrosis may be due to the action of a number of proteases. Blood. 2005 Jun 1;105(11):4508-15. doi: 10.1182/blood-2004-08-3238. Epub 2005 Feb 10. PMID 15705794
- [Background] Phelan JT 2nd, Prchal JT. Clonality studies in cancer based on X chromosome inactivation phenomenon. Methods Mol Med. 2002;68:251-70. doi: 10.1385/1-59259-135-3:251. No abstract available. PMID 11901507
- [Background] Damps-Konstanska I, Konstanski Z, Jassem E. [Treatment of pulmonary hypertension]. Wiad Lek. 2007;60(11-12):545-9. Polish. PMID 18540180
- [Background] Cortelezzi A, Gritti G, Del Papa N, Pasquini MC, Calori R, Gianelli U, Cortiana M, Parati G, Onida F, Sozzi F, Vener C, Bianchi P, Deliliers GL. Pulmonary arterial hypertension in primary myelofibrosis is common and associated with an altered angiogenic status. Leukemia. 2008 Mar;22(3):646-9. doi: 10.1038/sj.leu.2404943. Epub 2007 Sep 13. No abstract available. PMID 17851555
- [Background] Halank M, Marx C, Baretton G, Muller KM, Ehninger G, Hoffken G. Severe pulmonary hypertension in chronic idiopathic myelofibrosis. Onkologie. 2004 Oct;27(5):472-4. doi: 10.1159/000080368. PMID 15585978